CLINICAL TRIAL: NCT00617175
Title: ADVANCE III: Avoid DeliVering TherApies for Non-sustained Arrhythmias in ICD PatiEnts III
Brief Title: Avoid DeliVering TherApies for Non-sustained Arrhythmias in ICD PatiEnts III
Acronym: ADVANCEIII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADVANCE III; ADVANCE III
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Heart Disease
Keywords: Implantable Cardiac Defibrillator; therapies reduction; Shocks; Quality of Life
MeSH Terms: conditions — Heart Diseases; Shock | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long NID (Experimental): Programming a number of 30 out of 40 intervals to detect (NID)ventricular arrhythmia
  Interventions: Device: Implantable Defibrillator
- Short NID (Active Comparator): Programming a number of 18 out of 24 intervals to detect (NID)ventricular arrhythmia
  Interventions: Device: Implantable Defibrillator

INTERVENTIONS:
Device: Implantable Defibrillator — Number of 30 out of 40 intervals to detect (NID)Fast Ventricular Tachycardia
  Arms: Long NID
Device: Implantable Defibrillator — number of 18 out of 24 intervals to detect (NID)Fast Ventricular Tachycardia
  Arms: Short NID

SUMMARY:
To demonstrate a reduction in the number of ventricular therapies (ATP and Shocks) delivered for treating spontaneous arrhythmia episodes with a fast cycle length (CL≤ 320ms) as a consequence of self-termination and better arrhythmia discrimination due to a greater number of R-R intervals necessary to detect ventricular events.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective is to demonstrate a 20% reduction of ventricular therapies (ATP and Shocks) delivered for treating spontaneous arrhythmia episodes with a fast cycle length (CL ≤ 320 ms) by choosing a number of 30 out of 40 intervals to detect (NID) compared to a NID of 18 out of 24 in subjects with either Class I or IIA indication for ICD implantation, regardless of cardiac resynchronization capabilities.

Secondary Objectives:

1. Evaluate the percent reduction in the number of shocks delivered per subject for treating spontaneous episodes with a fast cycle length (CL ≤ 320 ms) and for spontaneous ventricular episodes.
2. Evaluate the efficacy of ATP in successfully treating spontaneous ventricular episodes (CL: 200ms-320ms) for subjects in primary and secondary prevention in both arms of the study.
3. Evaluate acceleration rate or degeneration into VF of spontaneous episodes (CL of 200ms-320ms) due to ATP therapy in the two study arms.
4. Compare the likelihood of syncopal events associated with spontaneous episodes with a fast cycle length (CL ≤ 320 ms).
5. Describe the economic impact and the quality of life consequences.

ELIGIBILITY:
Inclusion Criteria:

* Either ICD or CRT+ICD indications (Class I-IIA) according to the current AHA / ACC / ESC guidelines.
* Previous implant of a Medtronic device including "ATP During Charging" feature for 15 days at the maximum.

Exclusion Criteria:

* ICD replacements and upgrading.
* Brugada Syndrome, Long QT and HCM patients
* Ventricular tachyarrhythmia associated with reversible cause.
* Other electrical implantable devices (Neurostimulators, etc.).
* Subject's life expectancy less than 1 year.
* Subject on heart transplant list which is expected in less than 1 year.
* Subject is <18 years of age, or the subject is under a minimum age that is required as defined by local law
* Women who are pregnant or women of childbearing potential who are not on a reliable form of birth control.
* Unwillingness or inability to provide written informed consent.
* Enrolment in, or intention to participate in, another clinical trial.
* Inaccessibility to come to the study center for the follow-up visits.
* Mechanical tricuspid valve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorg O. Schwab, MD, Study Chair — University of Bonn, Bonn, Germany; Maurizio Gasparini, MD, Principal Investigator — Humanitas Hospital, Milano Italy; Maurizio Lunati, MD, Principal Investigator — Niguarda Hospital, Milano, Italy; Bernd Lemke, MD, Principal Investigator — Klinikum Lüdenscheid, Lüdenscheid, Germany; João Sousa, MD, Principal Investigator — H. Santa Maria - Lisbon - Portugal; Andrzej Okreglicki, MD, Principal Investigator — University of Cape Town, Cape Town, South Africa; Angel Arenal, MD, Principal Investigator — Hospital Gregorio Marañón, Madrid, Spain; Maurits Wijffels, MD, Principal Investigator — St. Antonius hospital - NIEUWEGEIN, The Netherlands
Locations (91):
- Belgium (5):
  - Hopital St-Joseph, Gilly
  - CHU Brugmann, Laken
  - CHR La Citadelle Liege, Liège
  - CHR Namur, Namur
  - AZ Nikolaas, Sint-Niklaas
- Denmark (2):
  - KAS Gentofte, Hellerup
  - Odense Universitets Hospital, Odense
- Turku University Central Hospital, Turku, Finland
- France (8):
  - Hôpital Michalon- CHU Grenoble, Grenoble
  - CHU Nantes - Hôpital Guillaume et René Laënnec, Nantes
  - NCN Nantes, Nantes
  - Hopital de la Pitie Salpetriere, Paris
  - Centre Hospitalier de Pau, Pau
  - CHU Hôpital de Pontchaillou Rennes, Rennes
  - CH Rangueil Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (9):
  - RWTH Aachen, Aachen
  - University of Bonn, Bonn
  - Kardiologisches Zentrum an der Klinik Rotes Kreuz, Frankfurt am Main
  - SRH Wald-Klinikum Gera gGmbH, Gera
  - Universitätskliniken des Saarlandes, Homburg
  - Klinikum Lüdenscheid, Lüdenscheid
  - Klinikum Dorothea Christiane Erxleben Quedlinburg, Quedlinburg
  - Universität Rostock- Medizinische Fakultät, Rostock
  - Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
- Hungary (2):
  - Semmelweis University AOK, Budapest
  - Zala County Hospital, Zalaegerszeg
- Italy (26):
  - Presidio Ospedaliero di Venere, Carbonara, Bari
  - Azienda.Ospedaliera.G.M. Lancisi, Ancona
  - Azienda Ospedaliera G. Rummo, Benevento
  - Cliniche Gavazzeni, Bergamo
  - Stab. Ospedaliero Di Summa-Perrino - Brindisi, Brindisi
  - Casa di Cura Mater Domini, Castellanza
  - Ospedale Pugliese e Ciaccio, Catanzaro
  - A.O. Santa Croce e Carle, Cuneo
  - Ente Ospedaliero Ospedali Galliera - Genova, Genova
  - Ospedale Maggiore di Lodi, Lodi
  - Istituto Ca' Granda-Niguarda, Milan
  - San Carlo Borromeo, Milan
  - Nuovo Osp. Civile S. Agostino, Modena
  - P.O. di Montebelluna, Montebelluna
  - Ospedale S. Giacomo, Novi Ligure
  - Policlinico S. Matteo, Pavia
  - Osp. S. Maria degli Angeli - Pordenone, Pordenone
  - Ospedale Misericordia e Dolce, Prato
  - Azienda Complesso Ospedaliero San Filippo Neri, Roma
  - Ospedale Sandro Pertini, Roma
  - Ospedale Sant Eugenio, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Osp. S. Giovanni di Dio e Ruggi dAragona, Salerno
  - AZ. Osp. Ordine Mauriziano, Torino
  - A.O. S.Maria della Misericordia, Udine
  - ULSS N.6 S. Bortolo - Vicenza, Vicenza
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
- Zoz Mswia, Bialystok, Poland
- Portugal (4):
  - Hospital Garcia Orta, SA, Almada
  - Hospital de Santa Maria, Lisbon
  - Hospital de Santa Marta, Lisbon
  - Hospital Geral de Santo António, Porto
- Tyumen Cardiology Center, Tyumen, Russia
- Saudi Arabia (2):
  - King Fahd Armed Forces Hospital, Jeddah
  - King Khalid Univ. Hospital - King Saud University, Riyadh
- South Africa (7):
  - Bloemfontein Medi-Clinic, Bloemfontein
  - Christiaan Barnard Memorial Hospital, Cape Town
  - University of Cape Town - Groote Schuur Hospital, Cape Town
  - Vincent Pallotti Hospital, Cape Town
  - Milpark Hospital, Johannesburg
  - Sunninghill Hospital, Johannesburg
  - UNITAS Hospital, Pretoria
- Spain (21):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de Basurto - Bilbao, Bilbao
  - Hospital General Yagüe, Burgos
  - Hospital General San Pedro de Alcantara, Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - H. Ramón y Cajal, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico de Malaga - Virgen de la Victoria, Málaga
  - Hospital Universitario Son Dureta, Palma Mallorca
  - Hospital Universitario de San Juan, Sant Joan d'Alacant
  - Hospital Ntra. Sra. de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Virgen de La Salud, Toledo
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Chuvi-Xeral-Cíes, Vigo
  - Hospital de Txagorritxu, Vitoria-Gasteiz

REFERENCES:
- [Derived] Landolina M, Boriani G, Biffi M, Cattafi G, Capucci A, Dello Russo A, Facchin D, Rordorf R, Sagone A, Del Greco M, Morani G, Nicolis D, Meloni S, Grammatico A, Gasparini M. Determinants of worse prognosis in patients with cardiac resynchronization therapy defibrillators. Are ventricular arrhythmias an adjunctive risk factor? J Cardiovasc Med (Hagerstown). 2022 Jan 1;23(1):42-48. doi: 10.2459/JCM.0000000000001236. PMID 34392257
- [Derived] Gasparini M, Kloppe A, Lunati M, Varma N, Martinez-Ferrer JB, Hersi A, Gulaj M, Wijffels MCEF, Arenal A, Mangoni di Santo Stefano L, Proclemer A. Sex differences in implantable cardiac defibrillator therapy according to arrhythmia detection times. Heart. 2020 Apr;106(7):520-526. doi: 10.1136/heartjnl-2019-315650. Epub 2019 Dec 11. PMID 31826936
- [Derived] Gasparini M, Lunati MG, Proclemer A, Arenal A, Kloppe A, Martinez Ferrer JB, Hersi AS, Gulaj M, Wijffels MCE, Santi E, Manotta L, Varma N. Long Detection Programming in Single-Chamber Defibrillators Reduces Unnecessary Therapies and Mortality: The ADVANCE III Trial. JACC Clin Electrophysiol. 2017 Nov;3(11):1275-1282. doi: 10.1016/j.jacep.2017.05.001. Epub 2017 May 31. PMID 29759624
- [Derived] Gasparini M, Kloppe A, Lunati M, Anselme F, Landolina M, Martinez-Ferrer JB, Proclemer A, Morani G, Biffi M, Ricci R, Rordorf R, Mangoni L, Manotta L, Grammatico A, Leyva F, Boriani G. Atrioventricular junction ablation in patients with atrial fibrillation treated with cardiac resynchronization therapy: positive impact on ventricular arrhythmias, implantable cardioverter-defibrillator therapies and hospitalizations. Eur J Heart Fail. 2018 Oct;20(10):1472-1481. doi: 10.1002/ejhf.1117. Epub 2017 Dec 18. PMID 29251799
- [Derived] Kloppe A, Proclemer A, Arenal A, Lunati M, Martinez Ferrer JB, Hersi A, Gulaj M, Wijffels MC, Santi E, Manotta L, Mangoni L, Gasparini M. Efficacy of long detection interval implantable cardioverter-defibrillator settings in secondary prevention population: data from the Avoid Delivering Therapies for Nonsustained Arrhythmias in ICD Patients III (ADVANCE III) trial. Circulation. 2014 Jul 22;130(4):308-14. doi: 10.1161/CIRCULATIONAHA.114.009468. Epub 2014 May 16. PMID 24838360
- [Derived] Gasparini M, Proclemer A, Klersy C, Kloppe A, Lunati M, Ferrer JB, Hersi A, Gulaj M, Wijfels MC, Santi E, Manotta L, Arenal A. Effect of long-detection interval vs standard-detection interval for implantable cardioverter-defibrillators on antitachycardia pacing and shock delivery: the ADVANCE III randomized clinical trial. JAMA. 2013 May 8;309(18):1903-11. doi: 10.1001/jama.2013.4598. PMID 23652522
- [Derived] Schwab JO, Gasparini M, Lunati M, Proclemer A, Kaup B, Santi E, Ligorio G, Klersy C, DE Sousa J, Okreglicki A, Arenal A, Wijffels M, Lemke B. Avoid delivering therapies for nonsustained fast ventricular tachyarrhythmia in patients with implantable cardioverter/defibrillator: the ADVANCE III Trial. J Cardiovasc Electrophysiol. 2009 Jun;20(6):663-6. doi: 10.1111/j.1540-8167.2008.01415.x. Epub 2009 Jan 9. PMID 19175450

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short NID | Long NID
Started | 954 | 948
Completed | 954 | 948
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short NID | Long NID | Total
Number analyzed (Participants) | 954 | 948 | 1902
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 391 | 390 | 781
  >=65 years | 563 | 558 | 1121
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (11.1) | 65.4 (11.0) | 65.47 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 153 | 304
  Male | 803 | 795 | 1598
Region of Enrollment [Number; unit: participants]
  Germany | 52 | 60 | 112
  Spain | 196 | 196 | 392
  Italy | 448 | 429 | 877
  Hungary | 11 | 9 | 20
  Netherlands | 25 | 23 | 48
  Belgium | 18 | 22 | 40
  France | 61 | 62 | 123
  Russian Federation | 9 | 18 | 27
  Saudi Arabia | 45 | 45 | 90
  Denmark | 9 | 14 | 23
  Finland | 3 | 2 | 5
  South Africa | 32 | 24 | 56
  Poland | 22 | 14 | 36
  Portugal | 23 | 30 | 53

OUTCOME MEASURES:

1. Primary Outcome: For the Primary Endpoint the Reduction of Ventricular Therapies (ATP and Shocks) Delivered for Treating Fast Spontaneous Arrhythmia Episodes Was Measured.
Description: for each patient, the exposure time was calculated as the period between randomization and until study completion or exit whichever occured first. Exposure times for all patients were then summed.
  The rate of therapies was calculated as the sum of all therapies delivered in the study (for each arm) over the sum of exposure times * 100.
Time Frame: From enrollment to study completion or exit whichever occured first
Population: For the primary endpoint analysis, only patients with at least a device data record were considered.
Measure: Number (95% Confidence Interval); unit: rate of therapies per 100 patient-years
Groups:
- NID 18/24: standard number of interval to detect ventricular arrhythmias
- NID 30/40: Prolonged number of interval to detect ventricular arrhythmias
Arm/Group | NID 18/24 | NID 30/40
Number analyzed (Participants) | 891 | 876
rate of therapies per 100 patient-years | 67.1 [61.7 to 72.9] | 41.9 [27.6 to 46.5]
Statistical Analysis 1: Comparison: NID 18/24 vs NID 30/40; Test type: Superiority or Other; p < 0.001, Negative binomial regression

2. Secondary Outcome: Evaluate the Percent Reduction in the Number of Shocks Delivered Per Subject for Treating Spontaneous Episodes With a Fast Cycle Length (CL < 320 ms) and for Spontaneous Ventricular Episodes.
Time Frame: end of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events collection started at day 0 after enrollment until study completion or exit whichever occured first.
Arm/Group | Short NID | Long NID
Serious Adverse Events (participants affected / at risk) | 300/954 | 258/948
Other Adverse Events (participants affected / at risk) | 0/954 | 0/948
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short NID (N=954) | Long NID (N=948)
Thromboembolic Events (Blood and lymphatic system disorders) | 16 | 8
Lead Dislodgment (Cardiac disorders) | 27 | 20
Worsening heart failure (Cardiac disorders) | 95 | 83
System Dysfunction (Cardiac disorders) | 1 | 1
Inappropriate Tachyarrhythmia Therapy (Cardiac disorders) | 7 | 5
Renal Failure (Renal and urinary disorders) | 10 | 8
Pocket Hematoma (Surgical and medical procedures) | 3 | 6
Post Surgical Infection (Surgical and medical procedures) | 5 | 3
Acute Myocardial Infarction (Cardiac disorders) | 9 | 11
Coronary Artery disease (Cardiac disorders) | 7 | 4
Elevated Threshold (Cardiac disorders) | 4 | 1
All cause syncope (Cardiac disorders) | 9 | 15
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Cardiogenic shock (Cardiac disorders) | 3 | 3
Ventricular Arrhythmia (Cardiac disorders) | 24 | 22
epicardial LV implant (Surgical and medical procedures) | 0 | 1
Pericardial Effusion (Surgical and medical procedures) | 1 | 2
Atrial Arrhthmias (Cardiac disorders) | 22 | 15
Pocket Infection (Surgical and medical procedures) | 11 | 17
Angina (Cardiac disorders) | 6 | 5
Extracardiac Stimulation (Cardiac disorders) | 2 | 3
Pneumothorax (Surgical and medical procedures) | 1 | 1
Dyspnea (Cardiac disorders) | 2 | 4
Neoplasia (General disorders) | 19 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Device migration (Surgical and medical procedures) | 1 | 3
hypotension (Blood and lymphatic system disorders) | 1 | 1
Hypertension (Blood and lymphatic system disorders) | 1 | 1
bradycardia (Cardiac disorders) | 1 | 0
Musculoskeletal diseases (Musculoskeletal and connective tissue disorders) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less